CLINICAL TRIAL: NCT02587845
Title: Use of Tranexamic Acid(TNA) in Preventing Blood Loss During and After Total Hip Arthroplasty
Brief Title: Use of Transexamic Acid in Hip Replacement
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Youn-Soo Park, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2014-01-129
Record Dates: First submitted 2014-04-24; First posted 2015-10-27 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Bleeding; Transfusion Related Complication
Keywords: total hip arthroplasty; transexamic acid
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IV group (Active Comparator): Intravenous tranexamic acid injection Group IV tranexamic acid group were administered intravenous 10 mg/kg dose of TXA after closing the ITB.
  Interventions: Drug: Tranexamic Acid (IV)
- Topical group (Experimental): Intra-articular tranexamic acid injection Group Topical tranexamic acid group were administered 2.0 g TXA in 100 ml of normal saline into the hemovac line after closing the ITB.
  Interventions: Drug: Tranexamic Acid (Topical)

INTERVENTIONS:
Drug: Tranexamic Acid (IV) — IV tranexamic acid group were administered intravenous 10 mg/kg dose of TXA after closing the ITB.
  Other Names: TXA
  Arms: IV group
Drug: Tranexamic Acid (Topical) — Topical tranexamic acid group were administered 2.0 g TXA in 100 ml of normal saline into the hemovac line after closing the ITB.
  Other Names: TXA
  Arms: Topical group

SUMMARY:
Studies have shown that tranexamic acid reduces blood loss and transfusion need in patients undergoing total hip arthroplasty. However, no to date, no study has been large enough to determine definitively whether the drug is safe and effective. The present study was designed to verify noninferior efficacy and safety of topical intra-articular TXA compared with intravenous TXA in primary THA.

DETAILED DESCRIPTION:
Treatment of choice for osteoarthritis of the hip, developmental dysplasia of the hip, and osteonecrosis of the femoral head in older patients. In association with the investigators aging society, the number of patients who will need THA may increase significantly in the next few years [1]. However, in THA, considerable blood loss remains a major problem, which can lead to a need for allogeneic blood transfusion. Such transfusion of allogeneic erythrocytes is not free of adverse events and has been associated with transmission of infectious diseases, increased postoperative bacterial infection, immune sensitization, transfusion-related acute lung injury, intravascular hemolysis, transfusion-induced coagulopathy, renal failure, admission to intensive care, and even death. Several effective interventions have been developed to reduce blood loss and postoperative transfusion rates, such as preoperative autologous donation, cell salvage, controlled hypotension, regional anesthesia, and the use of erythropoietin and antifibrinolytics. The antifibrinolytics include aprotinin, tranexamic acid (TXA), and ε-aminocaproic acid, which have different mechanisms of action [8]. TXA is a synthetic derivative of the amino acid lysine and a competitive inhibitor of plasminogen activation, and thus interferes with fibrinolysis. Compared with other antifibrinolytic drugs, TXA is cheaper and safer than aprotinin and more potent than the others. Numerous studies have evaluated the use of antifibrinolytics in orthopedic surgery and have shown them to be effective in reducing blood loss. However, the available clinical trials and meta-analyses lack sufficient statistical power to determine the effectiveness of antifibrinolytic agents in total hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral primary THA
* Diagnosis - not fracture, elective surgery
* Revision THA

Exclusion Criteria:

* Known allergy to TNA
* Acquired or congenital coagulopathy
* Current anticoagulation therapy
* Preoperative hepatic or renal dysfunction
* Severe ischemic heart disease (Serious cardiac or respiratory disease)
* A history of thromboembolic disease
* Refusal of blood products
* Pregnancy or breastfeeding

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Bleeding | intraoperatively
  Surgical bleeding

SECONDARY OUTCOMES:
Total Transfusion | 5days after surgery
  Allogenic transfusion

OTHER OUTCOMES:
Operation time | intraoperatively
  surgical time

CONTACTS AND LOCATIONS:
Overall Officials: Youn Soo Park, MD, Study Director — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea